CLINICAL TRIAL: NCT05044026
Title: A Prospective, Two-arm, Non Interventional Study of JAKAVI® (Ruxolitinib) in Patients With Myelofibrosis
Brief Title: A Prospective, Two-arm, Non-interventional Study of JAKAVI® (Ruxolitinib) in Patients With Myelofibrosis
Acronym: JAKoMo
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424ADE05
Record Dates: First submitted 2021-09-06; First posted 2021-09-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis
Keywords: Primary Myelofibrosis; PMF; post-polycythemia vera myelofibrosis; PPV MF; post-essential thrombocythemia myelofibrosis; post ET MF; Ruxolitinib; Jakavi
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm A: JAK inhibitor naive: JAK-inhibitor-naive patients, treatment start with ruxolitinib less than 14 days prior to the baseline visit
  Interventions: Other: Jakavi
- Arm B: Pretreated patients: Patients pretreated with a JAK-inhibitor for more than 14 days prior to the baseline visit
  Interventions: Other: Jakavi

INTERVENTIONS:
Other: Jakavi — Prospective observational study. There is no treatment allocation. Patients administered Jakavi by prescription and administered according to the SmPC.
  Other Names: Ruxolitinib

SUMMARY:
This was a prospective, two-arm, non-interventional study of JAKAVI® (Ruxolitinib) in patients with myelofibrosis

DETAILED DESCRIPTION:
The purpose of this NIS was to gather data from the daily clinical practice of the Jakavi®-treatment in a broad patient population. In order to evaluate the direct effect of Jakavi®, only JAK inhibitor naive patients were documented in the first study arm; patients pretreated with JAK inhibitors were documented in the second study arm to evaluate the long-term efficacy of Jakavi® in this subpopulation.

The documentation of all patients was carried out prospectively and began after the baseline visit. The medical decision on which therapeutic and diagnostic measures to take was made solely by the responsible physician. The observational period per patient was 36 months. The visit schedule after the baseline visit was set by the responsible physician according to standard clinical care, the clinical condition of the respective patients and the SmPC.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with Primary Myelofibrosis (PMF), post-Polycythemia Vera-Myelofibrosis (PPV-MF), or post-Essential Thrombocythemia-Myelofibrosis (post-ET-MF), for whom Jakavi® therapy is indicated.
* Patients that were informed about all aspects of this NIS and provided written informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (PPV-MF), or post-essential thrombocythemia Myelofibrosis (PET-MF), for whom Jakavi® therapy is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 1012 (Actual)
Dates: Start 2012-09-20 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 36 months
  Evaluation of all occurring adverse events, serious adverse events and serious and non-serious adverse drug reactions
Spleen size (or volume) reduction | Up to 36 months
  Spleen size (or volume) reduction was measured by palpation
Eastern Cooperative Oncology Group (ECOG) performance status | Up to 36 months
  The ECOG performance status is a scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  The grade ranges from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead).
Change in the number of patients with constitutional symptoms | Up to 36 months
  Number of patients with change in constitutional symptoms was collected
Assessment of the Quality of Life (QoL) - Myeloproliferative Neoplasm - Symptom Assessment Form (MPN-SAF) | Baseline, month 1, month 3, month 6, month 12, month 24 and month 36
  The MPN-SAF questionnaire contains important questions that cover MF-specific symptoms whose analysis is part of the standard of care. It includes disease related symptoms each scored from 0 (absent) to 10 (worst imaginable). Total Scores range from 0-100, with higher scores indicating a greater number of symptoms and severity.
Assessment of the Quality of Life (QoL) - Short Form-36 (SF-36) | Baseline month 6, month 12, month 24 and month 36
  This questionnaire consists of questions measuring physical function, physical role limitation, pain, general health, vitality, social function, emotional role limitations, and mental health status. The scores that can be obtained from the scale vary between 0 and 100 and the increase in the scores indicates that the quality of life is high.
Overall survival | Up to 36 months
  Overall survival for JAK inhibitor naive and pretreated patients
Ruxolitinib start and end dose | Up to 36 months
  Ruxolitinib start and end dose was collected
Therapy discontinuation and dose adjustments | Up to 36 months
  Number of participants with therapy discontinuation and dose adjustments was collected
Number of patients with co-morbidities | Up to 36 months
  Number of patients with co-morbidities was collected
Blood transfusion dependency | Up to 36 months
  Number of patients with blood transfusion dependency was collected
Number of patients with concomitant medications | Up to 36 months
  Number of patients with concomitant medications prescribed for myelofibrosis therapy and for the management of side effects was collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koschmieder S, Isfort S, Schulte C, Jacobasch L, Geer T, Reiser M, Koenigsmann M, Heinrich B, Wehmeyer J, von der Heyde E, Tesch H, Groschl B, Bachhuber P, Grosser S, Koehler M, Pahl HL. Final Results From a Large, Non-Interventional, Phase 4 Study of Ruxolitinib for the Treatment of Myelofibrosis in Clinical Routine. Eur J Haematol. 2025 Oct;115(4):380-390. doi: 10.1111/ejh.70005. Epub 2025 Jul 6. PMID 40619737
- [Derived] Koschmieder S, Isfort S, Schulte C, Jacobasch L, Geer T, Reiser M, Koenigsmann M, Heinrich B, Wehmeyer J, von der Heyde E, Tesch H, Groschl B, Bachhuber P, Grosser S, Pahl HL. Real-world analysis of ruxolitinib in myelofibrosis: interim results focusing on patients who were naive to JAK inhibitor therapy treated within the JAKoMo non-interventional, phase IV trial. Ann Hematol. 2023 Dec;102(12):3383-3399. doi: 10.1007/s00277-023-05458-1. Epub 2023 Oct 4. PMID 37792065
- See also: Results for CINC424ADE05 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18097